CLINICAL TRIAL: NCT03254758
Title: A Phase 1/2 Study of ADR-001 in Patients With Liver Cirrhosis
Brief Title: A Study of ADR-001 in Patients With Liver Cirrhosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rohto Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADR-001-01
Record Dates: First submitted 2017-08-03; First posted 2017-08-18 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Decompensated Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesenchymal stem cell (Experimental): Phase 1 Dose escalation : low Mid High Single administalation of ADR-001
  Phase 2 The recommended dose of ADR-001
  Interventions: Biological: Mesenchymal stem cell

INTERVENTIONS:
Biological: Mesenchymal stem cell — Phase1 The dose of AD-MSCs are escalated from low to mid and high step by step. Each administration is one time via intravenous infusion for one hour.
  Phase2 The recommended dose of ADR-001 is administrated once a week 4 times. The administration route and time is same method with Phase 1.

SUMMARY:
This is a first-in-human Phase1/2 study of ADR-001, adipose-derived mesenchymal stem cells (AD-MSCs). The safety and preliminary efficacy are evaluated in Phase 1 in patients with liver cirrhosis caused by Hepatitis C or Nonalcoholic Steatohepatitis and a recommended Phase 2 dose is determined by the evaluation. The exploratory efficacy and safety are investigated against the same target population in Phase 2.

DETAILED DESCRIPTION:
Patients with decompensated liver cirrhosis (Child-Pugh score; Grade B) caused by Hepatitis C or Nonalcoholic Steatohepatitis are enrolled to the study. In Phase 1, one of 3 doses of AD-MSCs is administered by 1 hour single intravenous infusion. Patients are hospitalized for 1 week and a recommended dose for Phase 2 is determined by the evaluation of the safety and efficacy. In Phase 2, patients with the same disease criteria are enrolled and dosed to investigate the exploratory efficacy and safety.

The safety and efficacy are evaluated until 24 weeks after dosing both in Phase 1 and Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 20 years of age
* Chronic hepatitis C or nonalcoholic steatohepatitis(NASH)
* Child-Pugh grade B liver cirrhosis
* ECOG Performance Status ≤ 2

Exclusion Criteria:

* Liver cirrhosis patients other than hepatitis C or NASH
* Malignant neoplasm (except hepatocellular carcinoma patients without recurrence more than 2 years)
* History of venous thrombosis or pulmonary embolism
* Serum creatinine ≥ 2 mg/dL or T-Bil ≥ 5.0 mg/dL
* Infection with hepatitis B, HIV, ATLV-1 or parvovirus B19
* Patients experienced transplantation or cell therapy
* Pregnancy or positive on pregnancy test
* Complications of significant heart disease, kidney disorder, or respiratory disease
* Drug or alcohol abuse

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Safety profile of ADR-001 including the incidence of adverse events (Phase 1) | 24 weeks
  Safety will be evaluated based on the medical review of adverse event reports and the results of clinical laboratory tests, vital sign, and physical examinations.
Improvement rate of Child-Pugh score (Phase 2) | 24 weeks
  Improvement rate of Child-Pugh score from the baseline will be evaluated.

SECONDARY OUTCOMES:
Change of liver function evaluated by Child-Pugh score (Phase 1) | 24 weeks
  Change of liver function from the baseline will be evaluated by Child-Pugh score.
Improvement rate of Child-Pugh score (Phase 1) | 24 weeks
  Improvement rate of Child-Pugh score from the baseline will be evaluated.
Improvement rate of Child-Pugh grade (Phase 1) | 24 weeks
  Improvement rate of Child-Pugh grade from the baseline will be evaluated.
Change of liver function evaluated by Child-Pugh score (Phase 2) | 24 weeks
  Change of liver function from the baseline will be evaluated by Child-Pugh score.
Improvement rate of Child-Pugh grade (Phase 2) | 24 weeks
  Improvement rate of Child-Pugh grade from the baseline will be evaluated.
Safety profile of ADR-001 including the incidence of adverse events (Phase 2) | 24 weeks
  Safety will be evaluated based on the medical review of adverse event reports and the results of clinical laboratory tests, vital sign, and physical examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Shuji Terai, MD, Principal Investigator — Niigata University Medical & Dental Hospital
Locations (2):
- Japan (2):
  - Niigata University Medical & Dental Hospital, Niigata
  - Nihon University Itabashi Hospital, Tokyo